CLINICAL TRIAL: NCT00493870
Title: Phase III Trial of TC Versus TAC in HER2-Negative Early Stage Breast Cancer Patients
Brief Title: TAC Versus TC for Adjuvant Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06090; 11271 (Other: Sanofi-Aventis)
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Results first posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TC (Experimental): docetaxel 75 mg/m2 and cyclophosphamide 600 mg/m2
  Interventions: Drug: Docetaxel; Drug: Cyclophosphamide
- TAC (Active Comparator): doxorubicin 50 mg/m2, cyclophosphamide 500 mg/m2 and docetaxel 75 mg/m2
  Interventions: Drug: Docetaxel; Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75 mg/m2 IV over 1 hour on Day 1 followed by cyclophosphamide
  Other Names: Taxotere
Drug: Doxorubicin — • Doxorubicin 50 mg/m2 IV push over 5-15 minutes via sidearm through a running IV line on Day 1, followed by cyclophosphamide 500 mg/m2 IV over 15-30 minutes on Day 1, followed by docetaxel 75 mg/m2 IV over 1 hour on Day 1. Administer pegfilgrastim 6 mg SC on Day 2 (or filgrastim 5 mcg/kg SC per standard of care).
  Other Names: Adriamycin
  Arms: TAC
Drug: Cyclophosphamide — 600 mg/m2 IV over 15-30 minutes on Day 1.
  Other Names: Cytoxan

SUMMARY:
The purpose of this research study is to find out what effects (good and bad) TC or TAC has on early stage HER2- breast cancer.

DETAILED DESCRIPTION:
Both TAC (docetaxel, doxorubicin, and cyclophosphamide) and TC (docetaxel and cyclophosphamide) are established adjuvant chemotherapy regimens for early stage breast cancer. TAC, however, due to the inclusion of the anthracycline doxorubicin, carries a high risk of hematologic and cardiotoxic adverse effects. Substantial evidence supports the concept that early stage HER2-negative breast cancers will benefit similarly from anthracycline-based adjuvant and non-anthracycline-based chemotherapy.

Further, approximately 0 to 9% of HER2-negative breast cancers have alterations in the TOP2A gene, which may predict for benefit from anthracycline-based chemotherapy.

We hypothesize that 6 cycles of TC versus 6 cycles of TAC will have similar efficacy in the treatment of early stage HER2-negative breast cancer and that TC will have less toxicity. If this hypothesis were upheld and the anthracycline doxorubicin could be eliminated from the regimen while obtaining similar efficacy in this population of patients, it would not only be an important advance in the understanding of the biology of cancer, but it would also be of significant clinical benefit to women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

A woman will be eligible for inclusion in this study if she meets all of the following criteria:

* Age >18 to <70 years old.
* Has known ER and PR status
* Has HER2 nonamplified disease, confirmed by FISH
* Has known menopausal status (see Section 7.3 for criteria)
* Has operable, histologically confirmed, Stage I, IIA, IIB, or IIIA, IIIB, or IIIC invasive carcinoma of the breast. Bilateral synchronous breast cancer is allowable provided that 1 primary meets the inclusion criteria.
* Meets 1 of the 3 following criteria:

  * T1-3N1-3M0 if ER positive or negative
  * T2-3N0M0 if ER positive or negative
  * T1N0M0 if ER and PR negative
* Has complete surgical resection of the primary breast tumor: either lumpectomy or mastectomy with sentinel lymph node biopsy or axillary dissection, with clear margins for both invasive and ductal carcinoma in situ (DCIS)
* Has had no prior chemotherapy unless >5 years ago
* Has an ECOG Performance Status (PS) 0-1
* Has laboratory values of: See protocol for specific details
* Has aspartate aminotransferase (AST) or alanine aminotransferase (ALT) and alkaline phosphatase (ALP) within the ranges shown below. In determining eligibility the more abnormal of the 2 values (AST or ALT) should be used. See protocol for specific details
* Has normal cardiac function as evidenced by a LVEF >50%, but WNL by institutional standard by multiple gated acquisition (MUGA) scan. An echocardiogram (ECHO) may be used if MUGA is not available, but the same modality must be used consistently throughout the study to evaluate LVEF. Ejection fraction as determined by ECHO must be WNL by institutional standard.
* Has no evidence of metastatic disease outside of breast by physical examination and chest x-ray. Other scans if done as needed by the patient (eg, bone scan; abdominal, chest CT; PET or PET/CT; ultrasound; or MRI should indicate no evidence of metastatic disease
* Has had baseline bilateral mammography
* It has been <84 days since the date of definitive surgery (eg, mastectomy or, in the case of a breast-sparing procedure, axillary dissection) with adequate wound healing, as determined by the Treating Physician
* Has a negative serum pregnancy test within 7 calendar days prior to registration (female patients of childbearing potential [not surgically sterilized and between menarche and 1 year postmenopause])
* If fertile, patient has agreed to use an acceptable method of birth control (barrier contraceptive only) to avoid pregnancy for the duration of the study and for a period of 3 months thereafter
* Has adequate tumor specimen available for FISH analysis of TOP2A status (See Appendix VI).
* Has signed a Patient Informed Consent Form
* Has signed a Patient Authorization Form

Exclusion Criteria:

A woman will be excluded from this study if she meets any of the following criteria:

* Has any evidence of metastatic disease following surgical resection of the primary tumor including: positive surgical margins, staging work-up, or physical examination suspicious for malignant disease
* Has T4 disease (ie, patients with fixed tumors, peau d'orange skin changes, skin ulcerations, or inflammatory changes)
* Has Stage IV breast cancer (M1 disease on TNM staging system)
* Has a history of severe hypersensitivity reaction to drugs formulated with polysorbate 80
* Has had neoadjuvant chemotherapy for this breast cancer
* Has ever had a myocardial infarction (MI) or has a history of heart failure, uncontrolled angina, severe uncontrolled arrhythmias, pericardial disease, or electrocardiographic evidence of acute ischemic changes
* Is receiving concurrent immunotherapy, hormonal therapy (eg, tamoxifen, hormone replacement therapy), or radiation therapy. Must discontinue prior to registering on the study.
* Is receiving concurrent investigational therapy or has received such therapy within the past 30 calendar days
* Has peripheral neuropathy >Grade 1
* Has had a major organ allograft or condition requiring chronic immunosuppression (ie, kidney, liver, lung, heart, bone marrow transplant, or autoimmune diseases). Patients who have received corneal transplants or cadaver skin or bone transplants are eligible.
* Has a serious uncontrolled intercurrent medical or psychiatric illness, including serious viral (including clinically defined AIDS), bacterial or fungal infection; or history of uncontrolled seizures, or diabetes, or CNS disorders deemed by the Treating Physician to be clinically significant, precluding informed consent
* Has active hepatitis B or hepatitis C with abnormal liver function tests (LFTs) or is known to be HIV positive
* Has a history of other malignancy within the last 5 years (except cured basal cell carcinoma of skin, carcinoma in situ of uterine cervix, DCIS, which could affect the diagnosis or assessment of any of the study drugs
* In an obese patient to whom the Treating Physician would not be comfortable administering full doses of study drugs as calculated by the BSA. Obese patients will be treated based on actual body weight. Obese patients treated with full doses based on actual BSA are eligible.
* Is pregnant or breastfeeding
* Is deemed unable to comply with requirements of study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1961 (Actual)
Dates: Start 2007-05-29 (Actual); Primary Completion 2015-05-31 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne L Blum, MD, Principal Investigator — US Oncology Research
Locations (94):
- United States (94):
  - Birmingham Hematology and Oncology, Birmingham, Alabama
  - Hematology Oncology Associates, Phoenix, Arizona
  - Northern AZ Hematology Oncology Associates-AOA, Sedona, Arizona
  - Arizona Oncology Associates DBA HOPE, Tucson, Arizona
  - Central Hematology Oncology Medical Group, Inc., Alhambra, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - St. Jude Hertiage Medical Group, Fullerton, California
  - Wilshire Oncology Medical Group, La Verne, California
  - Antelope Valley Cancer Center, Lancaster, California
  - Pacific Shores Medical Group, Long Beach, California
  - University of California-Los Angeles, Los Angeles, California
  - North Valley Hematology/Oncology Medical Group, Northridge, California
  - Ventura County Hematology-Oncology Specialist, Oxnard, California
  - SAMSUM Clinic, Santa Barbara, California
  - Santa Barabra Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Rocky Mountain Cancer Center-Rose, Denver, Colorado
  - Flordia Cancer Specialist, Fort Myers, Florida
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - Advanced Medical Specialist, Miami, Florida
  - Florida Cancer Institute, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - Suburban Hematology-Oncology Associates, PC, Lawrenceville, Georgia
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - Hematology Oncology Associates of IL, Chicago, Illinois
  - Cancer Care & Hematology Specialists of Chicagoland, Niles, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Hope Center, Terre Haute, Indiana
  - Kansas City Cancer Centers-Southwest, Overland Park, Kansas
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Alliance Hematology Oncology PA, Westminster, Maryland
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Arch Medical Services, Inc., St Louis, Missouri
  - Comprehensive Cancer Center of Nevada, Henderson, Nevada
  - Hematology-Oncology Associates of NNJ, P.A., Morristown, New Jersey
  - Southern New Mexico Cancer Center, Las Cruces, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - New York Oncology Hematology, P.C., Albany, New York
  - Interlakes Oncology Hematology, PC, Rochester, New York
  - Cancer Centers of North Carolina, Raleigh, North Carolina
  - Mahoning Valley Hematology Oncology Associates, Boardman, Ohio
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Medical Oncology Associates, Kingston, Pennsylvania
  - Rittenhouse Hematology/Oncology, Philadelphia, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Chattanooga Oncology & Hematology Associates, PC, Chattanooga, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Cancer Center-Abilene (South), Abilene, Texas
  - Texas Oncology, P.A.-Amarillo, Amarillo, Texas
  - Texas Cancer Center, Arlington, Texas
  - Texas Oncology Cancer Center, Austin, Texas
  - Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology -Bedford, Bedford, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology, Dallas, Texas
  - Methodist Charlton Cancer Ctr., Dallas, Texas
  - Texas Cancer Center, Denton, Texas
  - El Paso Cancer Treatment Ctr, El Paso, Texas
  - Texas Oncology, Fort Worth, Texas
  - Texas Oncology, Garland, Texas
  - Texas Oncology, P.A., Houston, Texas
  - Lake Vista Cancer Center, Lewisville, Texas
  - Longview Cancer Center, Longview, Texas
  - South Texas Cancer Center-McAllen, McAllen, Texas
  - Texas Cancer Center of Mesquite, Mesquite, Texas
  - Allison Cancer Center, Midland, Texas
  - Texas Oncology-Odessa, Odessa, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - South Texas Oncology and Hematology, P.A., San Antonio, Texas
  - San Antonio Tumor and Blood Clinic, San Antonio, Texas
  - HOAST-Medical Dr., San Antonio, Texas
  - Texas Cancer Center-Sherman, Sherman, Texas
  - Texas Oncology Cancer Center-Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology Cancer Care and Research, Waco, Texas
  - Texas Oncology PA, Webster, Texas
  - Texoma Cancer Center, Wichita Falls, Texas
  - Fairfax Northern VA Hem-Onc PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Onc and Hem Associates os SW VA, Inc., Salem, Virginia
  - Highline Medical Oncology, Burien, Washington
  - Pudget Sound Cancer Center-Edmonds, Edmonds, Washington
  - Columbia Basin Hematology and Oncology, Kennewick, Washington
  - Puget Sound Cancer Center-Seattle, Seattle, Washington
  - Cancer Care Northwest-South, Spokane, Washington
  - Northwest Cancer Specialists-Vancouver, Vancouver, Washington
  - Yakima Valley Mem Hosp/North Star Lodge, Yakima, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
  - Raleigh Regional Cancer Center, Beckley, West Virginia

REFERENCES:
- [Derived] Geyer CE Jr, Blum JL, Yothers G, Asmar L, Flynn PJ, Robert NJ, Hopkins JO, O'Shaughnessy JA, Rastogi P, Puhalla SL, Hilton CJ, Dang CT, Gomez HL, Vukelja SJ, Lyss AP, Paul D, Brufsky AM, Colangelo LH, Swain SM, Mamounas EP, Wolmark N. Long-Term Follow-Up of the Anthracyclines in Early Breast Cancer Trials (USOR 06-090, NSABP B-46-I/USOR 07132, and NSABP B-49 [NRG Oncology]). J Clin Oncol. 2024 Apr 20;42(12):1344-1349. doi: 10.1200/JCO.23.01428. Epub 2024 Feb 9. PMID 38335467

RESULTS

PARTICIPANT FLOW:
Groups:
- TC Arm: docetaxel 75 mg/m2 and cyclophosphamide 600 mg/m2
  Docetaxel: Docetaxel 75 mg/m2 IV over 1 hour on Day 1 plus Cyclophosphamide 600 mg/m2 IV over 15-30 minutes on Day 1 Q 21 day cycles X 6.
- TAC Arm: doxorubicin 50 mg/m2, cyclophosphamide 500 mg/m2 and docetaxel 75 mg/m2
  Docetaxel: Docetaxel 75 mg/m2 IV over 1 hour on Day 1 followed by cyclophosphamide
  Doxorubicin: • Doxorubicin 50 mg/m2 IV push over 5-15 minutes via sidearm through a running IV line on Day 1, plus cyclophosphamide 500 mg/m2 IV over 15-30 minutes on Day 1, plus docetaxel 75 mg/m2 IV over 1 hour on Day 1, followed by pegfilgrastim 6 mg SC (or filgrastim 5 mcg/kg SC) on Day 2 Q 21 day cycles X 6.
Period: Overall Study
Arm/Group | TC Arm | TAC Arm
Started | 981 | 980
Completed | 969 | 965
Not Completed | 12 | 15
Not completed — Lost to Follow-up | 12 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TC Arm | TAC Arm | Total
Number analyzed (Participants) | 969 | 965 | 1934
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (9.2) | 53.1 (8.9) | 53.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 969 | 965 | 1934
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 718 | 741 | 1459
  Hispanic | 141 | 97 | 238
  Black | 94 | 95 | 189
  Asian | 11 | 22 | 33
  Indian | 1 | 2 | 3
  Hawaiian | 0 | 2 | 2
  Other | 2 | 5 | 7
  Unknown | 2 | 1 | 3
Baseline Performance Status (ECOG) [Count of Participants; unit: Participants] — Score from 0-5 based on ECOG Performance Status scale:
  0: fully active, able to carry on all pre-disease performance without restriction
  1. : restricted in physically strenuous activity but able to walk & able to carry out work of a light nature
  2. : ambulatory & capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours
  3. : capable of only limited self-care, confined to bed or chair more than 50% of waking hours
  4. : completely disabled, cannot carry on any self-care, totally confined to bed or chair
  5. : dead
  Participants
    ECOG 0 | 860 | 857 | 1717
    ECOG 1 | 109 | 108 | 217
Stage [Count of Participants; unit: Participants] — Stages are as follows:
  I: The tumor in the breast is 20 millimeters (mm) or smaller in size at its widest area. This is a little less than an inch.
  II: The tumor is larger than 20 mm but not larger than 50 mm.
  III: The tumor is larger than 50 mm.
  Participants
    I | 136 | 124 | 260
    II | 705 | 716 | 1421
    III | 128 | 125 | 253
Hormone Receptor Status [Count of Participants; unit: Participants] — Hormone receptor-positive (or hormone-positive) breast cancer cells have either estrogen (ER) or progesterone (PR) receptors or both. These breast cancers can be treated with hormone therapy drugs that lower estrogen levels or block estrogen receptors.
  Participants
    Positive | 679 | 678 | 1357
    Negative | 290 | 287 | 577
Histology [Count of Participants; unit: Participants]
  Ductal | 811 | 789 | 1600
  Lobular | 87 | 100 | 187
  Mixed | 24 | 26 | 50
  Other | 47 | 48 | 95
  Unknown | 0 | 2 | 2
Tumor size [Mean (Standard Deviation); unit: cm] | 2.7 (1.5) | 2.6 (1.5) | 2.6 (1.5)
Positive Nodes [Count of Participants; unit: Participants] — Node-positive breast cancer means that cancer cells from the tumor in the breast have been found in the lymph nodes (sometimes called "glands") in the armpit area. The number of nodes involved are categorized here.
  Participants
    0 nodes | 358 | 339 | 697
    1-3 nodes | 455 | 480 | 935
    4-9 nodes | 116 | 111 | 227
    10+ nodes | 40 | 35 | 75
Grade [Count of Participants; unit: Participants]
  Well/Low | 100 | 119 | 219
  Moderately/Intermediate | 370 | 377 | 747
  Poorly/Undifferentiated | 470 | 431 | 901
  Unknown | 29 | 38 | 67
Menopausal Status [Count of Participants; unit: Participants]
  Peri | 41 | 42 | 83
  Post | 602 | 579 | 1181
  Pre | 324 | 343 | 667
  Unknown | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: 3-year Invasive Disease-free Survival (IDFS) Among Analyzed ITT Patients
Description: The primary objective of the study is to compare the 3-year invasive disease-free survival (IDFS) of adjuvant TC versus TAC as treatment for early stage HER2-negative breast cancer among analyzed ITT patients. ITT patients are all patients who were randomized, whether or not they followed protocol. IDFS, defined as the time from the date of randomization to local recurrence following mastectomy, invasive local recurrence in the ipsilateral breast following lumpectomy, regional recurrence, distant recurrence, invasive contralateral breast cancer, second primary cancer (other than squamous or basal cell carcinoma of the skin, melanoma in situ, carcinoma in situ of the cervix, colorectal carcinoma in situ, or lobular carcinoma in situ of the breast), or death from any cause prior to recurrence or second primary cancer. Patients who have not had any such event at the time of data analysis will be censored at the last date they were known to be event-free.
Time Frame: 3 years from randomization into study
Population: Analyzed ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TC Arm | TAC Arm
Number analyzed (Participants) | 969 | 965
percentage of participants | 91.1 [89.1 to 92.8] | 93.2 [91.3 to 94.6]
Statistical Analysis 1: Comparison: TC Arm vs TAC Arm; Test type: Other; p = 0.05, Log Rank

2. Primary Outcome: 3-year Invasive Disease-free Survival (IDFS) Among Per-protocol Patients
Description: The primary objective of the study is to compare the 3-year invasive disease-free survival (IDFS) of adjuvant TC versus TAC as treatment for early stage HER2-negative breast cancer among per-protocol patients. Per-protocol only includes those patients who were randomized and received treatment as outlined in the protocol.
Time Frame: 3 years from randomization into study
Population: Per-protocol patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TC Arm | TAC Arm
Number analyzed (Participants) | 950 | 934
percentage of participants | 91.3 [89.3 to 93.0] | 93.2 [91.3 to 94.7]

3. Secondary Outcome: 3-year DFS-DCIS, OS and RFI Among Analyzed ITT Patients
Description: To compare disease-free survival-ductal carcinoma in situ (DFS-DCIS),overall survival (OS) and recurrence free interval (RFI) of TC with TAC. DFS-DCIS, defined as the time from the date of randomization to local recurrence following mastectomy, local recurrence in the ipsilateral breast following lumpectomy (invasive or non-invasive), regional recurrence, distant recurrence, contralateral breast cancer (invasive or non-invasive), second primary cancer (other than squamous or basal cell carcinoma of the skin, melanoma in situ, carcinoma in situ of the cervix, colorectal carcinoma in situ, or lobular carcinoma in situ of the breast), or death from any cause prior to recurrence or second primary cancer. Patients who have not had any such event at the time of data analysis will be censored at the last date they were known to be event-free.
Time Frame: 3 years from randomization into study
Population: Analyzed ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TC Arm | TAC Arm
Number analyzed (Participants) | 969 | 965
percentage of participants
  3-year DFS-DCIS | 90.9 [88.8 to 92.6] | 93.0 [91.1 to 94.5]
  3-year OS | 96.8 [95.4 to 97.7] | 96.8 [95.5 to 97.8]
  3-year RFI | 91.9 [90.0 to 93.5] | 94.5 [92.8 to 95.9]

4. Secondary Outcome: 3-year DFS-DCIS, OS and RFI Among Per-protocol Patients.
Description: To compare disease-free survival-ductal carcinoma in situ (DFS-DCIS),overall survival (OS) and recurrence free interval (RFI) of TC with TAC among per protocol patients.
Time Frame: 3 years from randomization into study
Population: Analyzed per-protocol patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TC Arm | TAC Arm
Number analyzed (Participants) | 950 | 934
percentage of participants
  3-year DFS-DCIS | 91.1 [89.0 to 92.8] | 93.0 [91.1 to 94.5]
  3-year OS | 96.8 [95.5 to 97.8] | 96.8 [95.4 to 97.8]
  3-year RFI | 92.1 [90.2 to 93.7] | 94.5 [92.8 to 95.8]

5. Secondary Outcome: Number and Frequency of Participants by TOP2A Status by Study Treatment
Description: To evaluate the effectiveness of TC and TAC in TOP2A altered (amplified, deleted, or overexpressed at the protein level) early stage HER2-negative breast cancer
Time Frame: 10 years (from baseline to end of study participation)
Population: Analyzed ITT patients with TOP2A data
Measure: Count of Participants; unit: Participants
Arm/Group | TC Arm | TAC Arm
Number analyzed (Participants) | 624 | 631
Participants
  Amplification | 14 | 14
  Deletion | 131 | 128
  Normal | 479 | 489

6. Secondary Outcome: 3-year DFS Stratified by TOP2A Among TC Arm
Description: To evaluate DFS among TC in TOP2A altered (amplified, deleted, or overexpressed at the protein level) early stage HER2-negative breast cancer.
Time Frame: 3 years from randomization into study
Population: Analyzed ITT patients with TOP2A data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Amplification: TOP2A amplification subgroup in TC arm.
- Deletion: TOP2A deletion subgroup in TC arm.
- Normal: TOP2A normal subgroup in TC arm.
Arm/Group | Amplification | Deletion | Normal
Number analyzed (Participants) | 14 | 131 | 479
percentage of participants | 85.1 [52.3 to 96.1] | 82.8 [75.1 to 88.3] | 93.8 [91.2 to 95.6]

7. Secondary Outcome: 3-year DFS Stratified by TOP2A Among TAC Arm
Description: To evaluate DFS among TAC in TOP2A altered (amplified, deleted, or overexpressed at the protein level) early stage HER2-negative breast cancer.
Time Frame: 3 years from randomization into study
Population: Analyzed ITT patients with TOP2A data among TAC arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Amplification: TOP2A amplification subgroup in TAC arm.
- Deletion: TOP2A deletion subgroup in TAC arm.
- Normal: TOP2A normal subgroup in TAC arm.
Arm/Group | Amplification | Deletion | Normal
Number analyzed (Participants) | 14 | 128 | 489
percentage of participants | 100 [100 to 100] | 90.9 [84.2 to 94.9] | 93.2 [90.6 to 95.2]

ADVERSE EVENTS:
Time Frame: From Baseline to 30 days after last dose of study treatment, approximately 22 weeks. All-Cause Mortality was from baseline to end of study participation, approximately 10 years.
Arm/Group | TC Arm | TAC Arm
All-Cause Mortality (participants affected / at risk) | 110/969 | 88/965
Serious Adverse Events (participants affected / at risk) | 264/969 | 330/965
Other Adverse Events (participants affected / at risk) | 680/969 | 746/965
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TC Arm (N=969) | TAC Arm (N=965)
ALLERGY (Immune system disorders) | 2 (2) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 1 (1)
ASTHMA BRONCHIAL (Immune system disorders) | 0 (0) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
CIRCULATORY FAILURE (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HAEMOGLOBIN (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
LEUCOPENIA (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 8 (8) | 8 (8)
NEUTROPHIL COUNT (Blood and lymphatic system disorders) | 10 (10) | 18 (18)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
WBC INC (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 1 (1)
DEFECT CONDUCT INTRAVENTRICULAR (Cardiac disorders) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 1 (1)
TACHYCARDIA (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
ASYSTOLE (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC GENERAL - OTHER (SPECIFY) (Cardiac disorders) | 0 (0) | 1 (1)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 3 (3)
CONGESTIVE HEART FAILURE (Cardiac disorders) | 1 (1) | 1 (1)
HEART FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
HYPOTENSION (Cardiac disorders) | 4 (4) | 3 (3)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
CVA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
BROKEN CATHETER ON PORT-A-CATH (General disorders) | 0 (0) | 1 (1)
CHILLS (General disorders) | 1 (1) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 1 (1)
MALAISE (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1)
SHOCK (General disorders) | 0 (0) | 1 (1)
(General disorders) | 0 (0) | 1 (1)
WEAKNESS (General disorders) | 2 (2) | 0 (0)
SUDDEN DEATH (Investigations) | 0 (0) | 1 (1)
FOLLICULITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
BOWEL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
CAECITIS (Gastrointestinal disorders) | 0 (0) | 2 (2)
COLITIS (Gastrointestinal disorders) | 0 (0) | 4 (4)
DEHYDRATION (Gastrointestinal disorders) | 11 (11) | 18 (18)
DIARRHEA (Gastrointestinal disorders) | 11 (11) | 12 (12)
DIVERTICULITIS (Gastrointestinal disorders) | 0 (0) | 3 (3)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROENTERITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROESOPHAGEAL REFLUX (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI - OTHER (SPECIFY) (Gastrointestinal disorders) | 1 (1) | 1 (1)
GI HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
MUCOSITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 7 (7) | 10 (10)
PERFORATION COLON (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
STOOL BLOODY (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 8 (8) | 14 (14)
HEMATOMA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HEMORRHAGE, GI (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
LIVER FAILURE (Hepatobiliary disorders) | 1 (1) | 0 (0)
PANCREATITIS NOS (Hepatobiliary disorders) | 0 (0) | 1 (1)
ABSCESS (Infections and infestations) | 1 (1) | 4 (4)
ANAL INFECTION NOS (Infections and infestations) | 0 (0) | 1 (1)
BREAST INFECTION (Infections and infestations) | 2 (2) | 1 (1)
CELLULITIS (Infections and infestations) | 9 (9) | 5 (5)
CLOSTRIDIAL INFECTION NOS (Infections and infestations) | 1 (1) | 1 (1)
FEBRILE NEUTROPENIA (Infections and infestations) | 42 (42) | 44 (44)
FEVER (Infections and infestations) | 21 (21) | 13 (13)
INFECTION (DOCUMENTED CLINICALLY) (Infections and infestations) | 6 (6) | 4 (4)
INFECTION - OTHER (SPECIFY) (Infections and infestations) | 9 (9) | 10 (10)
INFECTION BACTERIAL (Infections and infestations) | 9 (9) | 8 (8)
INFECTION WITH NORMAL ANC (Infections and infestations) | 4 (4) | 0 (0)
INFECTION WITH UNKNOWN ANC (Infections and infestations) | 0 (0) | 1 (1)
INJECTION SITE INFECTION (Infections and infestations) | 1 (1) | 1 (1)
(Investigations) | 0 (0) | 4 (4)
OPPORTUNISITIC INFECTION (Infections and infestations) | 1 (1) | 1 (1)
PELVIC INFLAMMATION (Infections and infestations) | 0 (0) | 1 (1)
PERITONITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA NOS (Infections and infestations) | 1 (1) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1) | 3 (3)
SKIN INFECTION (Infections and infestations) | 3 (3) | 0 (0)
WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1)
EDEMA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
CONCENTRATION ABNORMAL (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
HYPOXEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DEVICE/PROSTHESIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
FRACTURE NOS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
CONFUSION (Nervous system disorders) | 1 (1) | 0 (0)
DEPRESSION (Nervous system disorders) | 0 (0) | 1 (1)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0)
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
MENTAL ACTIVITY DECREASED (Nervous system disorders) | 0 (0) | 1 (1)
MENTAL DISTRESS (Nervous system disorders) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Nervous system disorders) | 1 (1) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 1 (1)
PSYCHOSIS (Nervous system disorders) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1) | 2 (2)
SYNCOPE (Nervous system disorders) | 2 (2) | 3 (3)
SYNCOPE VASOVAGAL (Nervous system disorders) | 0 (0) | 1 (1)
VIOLENT (Nervous system disorders) | 0 (0) | 1 (1)
AMAUROSIS (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Investigations) | 7 (7) | 10 (10)
BACK PAIN (Investigations) | 3 (3) | 0 (0)
BONE PAIN (Investigations) | 1 (1) | 0 (0)
CHEST PAIN (Investigations) | 5 (5) | 4 (4)
HEADACHE (Investigations) | 0 (0) | 2 (2)
PAIN (Investigations) | 3 (3) | 7 (7)
PAIN PELVIC (Investigations) | 0 (0) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BREATH SHORTNESS (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
EMBOLISM PULMONARY (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
PULMONARY INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ANTIDIURETIC HORMONE DISORDER (Renal and urinary disorders) | 1 (1) | 0 (0)
BLADDER INFECTION (Renal and urinary disorders) | 2 (2) | 2 (2)
HEMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 3 (3)
SECONDARY MALIGNANCY (POSSIBLY RELATED TO CANCER TREATME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
MENORRHAGIA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
THROMBOSIS (Vascular disorders) | 1 (1) | 9 (9)
VASCULAR ACCESS NOS COMPLICATION (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TC Arm (N=969) | TAC Arm (N=965)
ANEMIA (Blood and lymphatic system disorders) | 164 (164) | 183 (183)
LEUCOPENIA (Blood and lymphatic system disorders) | 100 (100) | 92 (92)
NEUTROPENIA (Blood and lymphatic system disorders) | 294 (294) | 243 (243)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 18 (18) | 72 (72)
FATIGUE (General disorders) | 470 (470) | 498 (498)
ALOPECIA (Skin and subcutaneous tissue disorders) | 543 (543) | 538 (538)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 100 (100) | 58 (58)
RASH (Skin and subcutaneous tissue disorders) | 168 (168) | 94 (94)
HOT FLASHES (Endocrine disorders) | 95 (95) | 80 (80)
ANOREXIA (Gastrointestinal disorders) | 77 (77) | 107 (107)
CONSTIPATION (Gastrointestinal disorders) | 153 (153) | 175 (175)
DEHYDRATION (Gastrointestinal disorders) | 33 (33) | 85 (85)
DIARRHEA (Gastrointestinal disorders) | 251 (251) | 331 (331)
DYSGEUSIA (Gastrointestinal disorders) | 106 (106) | 127 (127)
GASTROESOPHAGEAL REFLUX (Gastrointestinal disorders) | 75 (75) | 97 (97)
MUCOSITIS (Gastrointestinal disorders) | 84 (84) | 94 (94)
NAUSEA (Gastrointestinal disorders) | 326 (326) | 413 (413)
STOMATITIS (Gastrointestinal disorders) | 69 (69) | 63 (63)
VOMITING (Gastrointestinal disorders) | 114 (114) | 164 (164)
FEVER (Infections and infestations) | 78 (78) | 80 (80)
INFECTION BACTERIAL (Infections and infestations) | 43 (43) | 50 (50)
INFECTION FUNGAL (Infections and infestations) | 31 (31) | 51 (51)
EDEMA (Blood and lymphatic system disorders) | 188 (188) | 142 (142)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 53 (53) | 56 (56)
ANXIETY (Nervous system disorders) | 63 (63) | 56 (56)
DEPRESSION (Nervous system disorders) | 59 (59) | 46 (46)
DIZZINESS (Nervous system disorders) | 42 (42) | 54 (54)
INSOMNIA (Nervous system disorders) | 102 (102) | 92 (92)
NEUROPATHY (Nervous system disorders) | 203 (203) | 171 (171)
EPIPHORA (Eye disorders) | 58 (58) | 61 (61)
ABDOMINAL PAIN (Investigations) | 56 (56) | 75 (75)
ARTHRALGIA (Investigations) | 128 (128) | 100 (100)
BACK PAIN (Investigations) | 52 (52) | 52 (52)
BONE PAIN (Investigations) | 113 (113) | 104 (104)
HEADACHE (Investigations) | 112 (112) | 112 (112)
MYALGIA (Investigations) | 144 (144) | 109 (109)
PAIN (Investigations) | 185 (185) | 139 (139)
BREATH SHORTNESS (Respiratory, thoracic and mediastinal disorders) | 65 (65) | 66 (66)
COUGH (Respiratory, thoracic and mediastinal disorders) | 76 (76) | 88 (88)
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 54 (54) | 37 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days